CLINICAL TRIAL: NCT06691516
Title: Radiographic Assessment Of The Accuracy Of 3D Ridge Augmentation In Anterior Mandible Using Computer Guided Autogenous Cortical Shell Technique Versus Free Hand Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Sayed Ibrahim Elballal, Dr.Ahmed Salah, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Computer guided cortical shell
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Bone Loss
Keywords: cortical shell , bone loss , computer guided
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guide cortical shell technique in anterior mandible 3d defect (Experimental): in study group there are bone harvesting guide and two fixation guides
  Interventions: Procedure: horizontal and vertical bone augmentation using computer guided cortical shell technique
- free hand cortical shell technique in anterior 3d defect (Active Comparator): in control group, the bone harvesting and shells fixation will done with free hand technique
  Interventions: Procedure: free hand cortical shell technique in anterior 3d defect

INTERVENTIONS:
Procedure: horizontal and vertical bone augmentation using computer guided cortical shell technique — Computer-guided cortical shell technique in anterior mandible 3d defect using bone harvesting guide and fixation guides
  Arms: computer guide cortical shell technique in anterior mandible 3d defect
Procedure: free hand cortical shell technique in anterior 3d defect — vertical and horizontal ridge augmentation in anterior mandible using free hand cortical shell technique
  Arms: free hand cortical shell technique in anterior 3d defect

SUMMARY:
* this study aims to evaluate accuracy of fixation of the bone shells by a calculated distance which is always a challenging step for inexperienced surgeons to fix a cortical shells at the ideal position in the conventional protocol.

the fixation guides used to make the shells precisely fixed at the proper position and angulation the problem is if it fixed with insufficient distance with proposed volume loss leads to totally insufficient volume gain for future implant placement

* also to evaluate the efficacy of the CAD/CAM surgical guide during chin harvesting (harvesting guide ) procedure in reducing the risk of anatomical structure damage (mental neve) and patient morbidity with more accuracy compared with the standard technique and preserve the roots of the lower anterior teeth or any fracture to the inferior border of the mandible also allow to harvest the bone shells from the suitable area with cancellous bone which prevent bad split of the bone shells this trial versus free hand conventional cortical shell bone technique both harvested from symphysis area (chin),
* also to evaluate thickness of implanted bone shells , the thickness should be enough to preserve the graft(autograft 50% and xenograft 50%) between the buccal and lingual bone shells
* also aims to evaluate the vertical and horizontal bone augmentation achieved at the anterior mandible using computer-guided cortical shell bone technique.

DETAILED DESCRIPTION:
this study aims to evaluate accuracy of fixation of the bone shells by a calculated distance which is always a challenging step for inexperienced surgeons to fix a cortical shells at the ideal position in the conventional protocol.

the fixation guides used to make the shells precisely fixed at the proper position and angulation the problem is if it fixed with insufficient distance with proposed volume loss leads to totally insufficient volume gain for future implant placement

* also to evaluate the efficacy of the CAD/CAM surgical guide during chin harvesting (harvesting guide ) procedure in reducing the risk of anatomical structure damage (mental neve) and patient morbidity with more accuracy compared with the standard technique and preserve the roots of the lower anterior teeth or any fracture to the inferior border of the mandible also allow to harvest the bone shells from the suitable area with cancellous bone which prevent bad split of the bone shells this trial versus free hand conventional cortical shell bone technique both harvested from symphysis area (chin),
* also to evaluate thickness of implanted bone shells , the thickness should be enough to preserve the graft(autograft 50% and xenograft 50%) between the buccal and lingual bone shells
* also aims to evaluate the vertical and horizontal bone augmentation achieved at the anterior mandible using computer-guided cortical shell bone technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 20-60 years. No sex predilection.

Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.

Edentulous anterior mandible with a horizontally deficient alveolar ridge that is less than 3mm in width and with a vertically defect at least 3mm in height.

The minimum number of missing teeth in the anterior mandible alveolar ridge is two adjacent teeth.

Exclusion Criteria:

* Intra-bony lesions (e.g., cysts) or infections (e.g., abscess) that may retard the osteotomy healing.

Previous grafting procedures in the edentulous area

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11-21 (Estimated); Primary Completion 2025-12-26 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of the implanted bone blocks | immediately post operative
  * depening on the superimposition between immediate postoperative CBCT scan over planning
  * the maximum thickness of the implanted bone blocks (mimics)

SECONDARY OUTCOMES:
bone gain vertical and horizontal | 6 months
  CBCT volumetric change of deficient alveolar ridge after augmentation